CLINICAL TRIAL: NCT00124345
Title: The Humidification During Noninvasive Mechanical Ventilation Delivered by Helmet
Brief Title: Medical Gas Humidification During Noninvasive Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Davide Chiumello, Policlinico Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1457
Record Dates: First submitted 2005-07-26; First posted 2005-07-27 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Respiration, Artificial; Critical Illness
Keywords: temperature; humidity; non invasive mechanical ventilation
MeSH Terms: conditions — Respiratory Aspiration; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: MR730

INTERVENTIONS:
Device: MR730 — humidity measurement inside the helmet by a capacitative hygrometer and evaluation of patients' comfort

SUMMARY:
In this study, the investigators aimed to study the role of medical gas humidification during noninvasive mechanical ventilation.

DETAILED DESCRIPTION:
The medical gases are usually dry and cold thus when they are used during invasive mechanical ventilation they must be conditioned. No data are present on the necessity to condition the medical gases during non invasive mechanical ventilation. In this study the investigators studied the humidity and the temperature of the medical gases with and without any conditioning during non invasive mechanical ventilation in a group of healthy subjects and critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients requiring non invasive mechanical ventilation

Exclusion Criteria:

* Comatose patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The level of temperature and humidity | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy